CLINICAL TRIAL: NCT03171545
Title: Enhancing the Cardiovascular Safety of Hemodialysis Care: A Cluster-Randomized, Comparative Effectiveness Trial of Multimodal Provider Education and Patient Activation Interventions (Dialysafe)
Brief Title: Enhancing the Cardiovascular Safety of Hemodialysis Care (Dialysafe)
Acronym: Dialysafe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of California, Irvine (Other); National Kidney Foundation, United States (Other); Fresenius Medical Care North America (Industry)
Responsible Party: Principal Investigator, Tiffany Veinot, Joan C. Durrance Collegiate Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HUM00125305; IHS-1503-27848 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Kidney Failure; End Stage Renal Disease; Hypotension; Cardiovascular Diseases; Patient Safety
Keywords: Peer Mentoring; Team Training; Checklist
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic; Hypotension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The study is a 2X2 factorial design, such that five facilities will get the provider education only; five will get the patient activation intervention only; five will get both interventions; and five will get no interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patient Activation (Experimental): This arm focuses on patients. It includes peer mentoring by trained End Stage Renal Disease (ESRD) patients. Mentors will hold 5 multimedia-aided meetings with other patients that include motivational interviewing and role modeling.
  Interventions: Behavioral: Patient Activation
- Provider Education (Experimental): This arm focuses on dialysis facility care teams. It includes team training, online education, and checklists.
  Interventions: Behavioral: Provider Education
- No Intervention (No Intervention): Patients in clinic receive usual care.
- Patient and Provider (Experimental): This arm includes both Patient Activation and Provider Education interventions
  Interventions: Behavioral: Patient Activation; Behavioral: Provider Education

INTERVENTIONS:
Behavioral: Patient Activation — Patients in clinics assigned to this group will be offered peer mentoring and digital resources.
  Arms: Patient Activation; Patient and Provider
Behavioral: Provider Education — Staff in clinics assigned to this group will receive team training and a checklist.
  Arms: Patient and Provider; Provider Education

SUMMARY:
The purpose of this study is reduce episodes of intradialytic hypotension, low blood pressure during a hemodialysis session, in patients with End Stage Renal Disease (ESRD). Recruitment will take place on the clinic level rather than the patient level.

DETAILED DESCRIPTION:
When a person's kidneys stop working, he or she has end-stage renal disease (ESRD). Individuals with ESRD cannot live without either dialysis therapy-in which a machine performs the functions of the kidneys-or a kidney transplant. Dialysis must remove fluid as well as toxins in the blood. People with ESRD have a high risk for death, and the usual cause is cardiovascular disease.

Most people in the United States who have ESRD get hemodialysis therapy in a clinic for four hours at a time, three times a week. The stability of hemodialysis sessions varies, and many sessions become unstable from low blood pressure and other complications. Unstable dialysis sessions can result in negative symptoms, like fatigue.

Dialysis instability is an important problem. Session instability is linked to injury to the heart and other organs. Patients who have unstable dialysis sessions are more likely to end up in the hospital or die than are those who have stable sessions. Session instability is preventable. The main causes of instability are removal of fluid from a patient too fast or removal of too much fluid. Session instability results from many factors: decisions made by patients, and decisions by healthcare providers.

Presently, the way to best improve the stability of dialysis is not clear. Dialysis clinics approach this problem differently, and there is variation among clinics in how often hemodialysis sessions become unstable.

In partnership with the National Kidney Foundation and Fresenius Medical Care North America, the investigators will test two interventions designed to increase the stability of patient dialysis. One intervention, multimodal provider education, focuses on dialysis facility care teams. It includes team training, online education, and a checklist. Another intervention, patient activation, focuses on patients. It includes peer mentoring by trained ESRD patients. Mentors will hold with other patients multimedia-aided meetings that include skills instruction and role modeling. These interventions have been successful in hospital care and in chronic disease care, and the investigators will adapt them to dialysis safety.

The investigators will then conduct a study in 20 dialysis facilities in different parts of the United States. Five facilities will get the provider education only; five will get the patient activation intervention only; five will get both interventions; and five will get no interventions. The investigators will test whether session stability improves in the facilities that get either intervention over the 48-week study period. This study is expected to clarify whether these interventions can make dialysis safer for ESRD patients. This will inform hemodialysis care providers on whether to pursue provider-focused or patient-focused safety interventions, or both. People on hemodialysis will also have information to help them decide whether to become engaged in their session stability, and the intervention will help them learn how to do so.

ELIGIBILITY:
Selection is at both the clinic level and individual patient level.

Clinic Inclusion Criteria:

* outpatient hemodialysis facilities
* at least 70 adult (>21 years old) patients to guarantee sample size

Clinic Exclusion Criteria:

* facilities involved in another study
* facilities in immediate jeopardy
* facilities with 1-star quality ratings
* facilities designated as COVID-19 isolation facilities

Individual Patient Exclusion Criteria:

* individual patients who are currently incarcerated
* individual patients who have poor cognition or cognitive impairment
* individual patients unable to comprehend the patient information sheet due to lack of facility in English or Spanish
* individual patients who have opted out of data collection

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1431 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-11-17 (Actual); Study Completion 2024-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Veinot, PhD, Principal Investigator — University of Michigan
Locations (1):
- Fresenius Kidney Care University Of Michigan - Ann Arbor, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veinot TC, Gillespie B, Argentina M, Bragg-Gresham J, Chatoth D, Collins Damron K, Heung M, Krein S, Wingard R, Zheng K, Saran R. Enhancing the Cardiovascular Safety of Hemodialysis Care Using Multimodal Provider Education and Patient Activation Interventions: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2023 Apr 20;12:e46187. doi: 10.2196/46187. PMID 37079365
- [Background] Veinot TC, Clarke PJ, Romero DM, Buis LR, Dillahunt TR, Vydiswaran VVG, Beals A, Brown L, Richards O, Williamson A, Antonio MG. Equitable Research PRAXIS: A Framework for Health Informatics Methods. Yearb Med Inform. 2022 Aug;31(1):307-316. doi: 10.1055/s-0042-1742542. Epub 2022 Dec 4. PMID 36463889
- [Background] Willis M, Brand Hein L, Hu Z, Saran R, Argentina M, Bragg-Gresham J, Krein SL, Gillespie B, Zheng K, Veinot TC. Usability Evaluation of a Tablet-Based Intervention to Prevent Intradialytic Hypotension in Dialysis Patients During In-Clinic Dialysis: Mixed Methods Study. JMIR Hum Factors. 2021 Jun 14;8(2):e26012. doi: 10.2196/26012. PMID 34121664
- [Background] Willis MA, Hein LB, Hu Z, Saran R, Argentina M, Bragg-Gresham J, Krein SL, Gillespie B, Zheng K, Veinot TC. Feeling better on hemodialysis: user-centered design requirements for promoting patient involvement in the prevention of treatment complications. J Am Med Inform Assoc. 2021 Jul 30;28(8):1612-1631. doi: 10.1093/jamia/ocab033. PMID 34117493
- [Background] Kuo PY, Saran R, Argentina M, Heung M, Bragg-Gresham J, Krein S, Gillespie BW, Zheng K, Veinot TC. Cramping, crashing, cannulating, and clotting: a qualitative study of patients' definitions of a "bad run" on hemodialysis. BMC Nephrol. 2020 Feb 27;21(1):67. doi: 10.1186/s12882-020-01726-8. PMID 32103726
- [Background] Kuo PY, Saran R, Argentina M, Heung M, Bragg-Gresham JL, Chatoth D, Gillespie B, Krein S, Wingard R, Zheng K, Veinot TC. Development of a checklist for the prevention of intradialytic hypotension in hemodialysis care: Design considerations based on activity theory. In: Proceedings of the 2019 CHI Conference on Human Factors in Computing Systems 2019 May 2 (pp. 1-14).

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Hemodialysis Facilities
Period: Baseline
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Started (12 week retrospective baseline; "not completed" if participants became ineligible for study between the enrollment period and start of intervention) | 382; 5 Hemodialysis Facilities | 346; 5 Hemodialysis Facilities | 410; 5 Hemodialysis Facilities | 293; 5 Hemodialysis Facilities
Completed | 377; 5 Hemodialysis Facilities | 342; 5 Hemodialysis Facilities | 401; 5 Hemodialysis Facilities | 286; 5 Hemodialysis Facilities
Not Completed | 5; 0 Hemodialysis Facilities | 4; 0 Hemodialysis Facilities | 9; 0 Hemodialysis Facilities | 7; 0 Hemodialysis Facilities
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Transferred out of clinic | 4 | 0 | 2 | 0
Not completed — Death | 1 | 2 | 1 | 5
Not completed — Recovered renal function | 0 | 0 | 1 | 0
Not completed — Received transplant | 0 | 0 | 1 | 0
Not completed — No longer receiving in-center hemodialysis | 0 | 2 | 3 | 0
Period: Intervention
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Started (24 week intervention period) | 377; 5 Hemodialysis Facilities | 342; 5 Hemodialysis Facilities | 401; 5 Hemodialysis Facilities | 286; 5 Hemodialysis Facilities
Completed | 323; 5 Hemodialysis Facilities | 307; 5 Hemodialysis Facilities | 348; 5 Hemodialysis Facilities | 247; 5 Hemodialysis Facilities
Not Completed | 54; 0 Hemodialysis Facilities | 35; 0 Hemodialysis Facilities | 53; 0 Hemodialysis Facilities | 39; 0 Hemodialysis Facilities
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 4
Not completed — Transferred out of clinic | 12 | 9 | 17 | 9
Not completed — Death | 26 | 16 | 29 | 14
Not completed — Received transplant | 7 | 5 | 3 | 6
Not completed — No longer receiving in-center hemodialysis | 7 | 4 | 4 | 6
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: Follow up
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Started (12 week follow up period) | 323; 5 Hemodialysis Facilities | 307; 5 Hemodialysis Facilities | 348; 5 Hemodialysis Facilities | 247; 5 Hemodialysis Facilities
Completed | 291; 5 Hemodialysis Facilities | 285; 5 Hemodialysis Facilities | 327; 5 Hemodialysis Facilities | 230; 5 Hemodialysis Facilities
Not Completed | 32; 0 Hemodialysis Facilities | 22; 0 Hemodialysis Facilities | 21; 0 Hemodialysis Facilities | 17; 0 Hemodialysis Facilities
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Transferred out of clinic | 4 | 4 | 12 | 7
Not completed — Death | 18 | 12 | 5 | 8
Not completed — Received transplant | 4 | 1 | 0 | 1
Not completed — No longer receiving in-center hemodialysis | 4 | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: These are all participants who were analyzed for baseline data, i.e. all enrolled participants regardless of how long they were enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider | Total
Number analyzed (Participants) | 382 | 346 | 410 | 293 | 1431
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.45 (13.92) | 63.58 (14.72) | 59.90 (13.36) | 61.66 (14.70) | 62.63 (14.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 154 | 162 | 115 | 594
  Male | 219 | 192 | 248 | 178 | 837
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 6 | 6 | 9 | 3 | 24
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 0 | 0 | 5
  Black or African American | 115 | 91 | 233 | 130 | 569
  White | 252 | 233 | 157 | 147 | 789
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 14 | 10 | 13 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71 | 68 | 38 | 32 | 209
  Not Hispanic or Latino | 307 | 265 | 353 | 245 | 1170
  Unknown or Not Reported | 4 | 13 | 19 | 16 | 52
Dialysis Session Stability [Mean (Standard Deviation); unit: Proportion of sessions] — Systolic blood pressure (SBP) falling below 100 mmHg (using lowest SBP during session) if starting SBP ≥100.
  Proportion of sessions | 0.197 (0.215) | 0.198 (0.212) | 0.175 (0.206) | 0.177 (0.213) | 0.187 (0.212)

OUTCOME MEASURES:

1. Secondary Outcome: Fluid Adherence
Description: Measured by interdialytic weight gain (in Kilograms), which is the weight gained between dialysis sessions (presented as average throughout 24 week intervention period)
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Number analyzed (Participants) | 377 | 342 | 401 | 286
Kg | 2.12 (0.87) | 2.18 (1.18) | 2.35 (0.93) | 2.34 (1.01)

2. Secondary Outcome: Dialysis Adherence - Average Weekly Minutes Missed Over Intervention Period
Description: Measured as the average number of minutes of prescribed dialysis time missed per week during intervention period (number of prescribed minutes-number of actual minutes/24 week intervention period).
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: average weekly minutes
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Number analyzed (Participants) | 377 | 342 | 401 | 286
average weekly minutes | 5.23 (13.48) | 4.21 (9.05) | 5.28 (10.58) | 4.89 (11.69)

3. Secondary Outcome: Dialysis Adherence - Average Weekly Sessions Missed During Intervention Period
Description: Measured as the average number of missed sessions per week during the intervention period (number of prescribed sessions-number of actual sessions/24 week intervention period).
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: average proportion of sessions missed
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Number analyzed (Participants) | 377 | 342 | 401 | 286
average proportion of sessions missed | 0.004 (0.008) | 0.008 (0.041) | 0.028 (0.061) | 0.032 (0.077)

4. Secondary Outcome: Patient Symptoms - Post-dialysis Recovery Time
Description: Measured at midweek session as patient recovery time after dialysis, reported on a survey item on an ordinal scale from "within minutes" to "did not recover before the next scheduled dialysis session." Responses grouped into three categories for analysis: "did not recover," "recovered before reaching home," and "recovered on same day of treatment." Sessions categorized as "recovered before reaching home" used for comparison between study arms.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Proportion session recovery before home
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Number analyzed (Participants) | 377 | 342 | 401 | 286
Proportion session recovery before home | 0.141 (0.106) | 0.181 (0.091) | 0.178 (0.091) | 0.158 (0.108)

5. Secondary Outcome: Patient Symptoms - Symptom Burden
Description: Measured as the total number symptoms reported by the patient at each session (each symptom treated as one, then added to create total symptoms).
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Average symptoms reported per session
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Number analyzed (Participants) | 377 | 342 | 401 | 286
Average symptoms reported per session | 0.045 (0.095) | 0.069 (0.154) | 0.051 (0.123) | 0.063 (0.133)

6. Secondary Outcome: Quality of Life-KDQOL - MCS
Description: Total score measured by adding responses on the Kidney Disease Quality of Life survey (KDQOLTM-36 Version 1). MCS (mental component summary) subscale ranges from 5.8 - 69.9; higher scores represent better functioning.
Time Frame: post-intervention survey
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Number analyzed (Participants) | 162 | 125 | 158 | 132
Score | 53.85 (8.73) | 52.62 (10.16) | 54.58 (8.30) | 54.89 (8.67)

7. Secondary Outcome: Quality of Life-KDQOL - PCS
Description: Total score measured by adding responses on the Kidney Disease Quality of Life survey (KDQOLTM-36 Version 1). PCS (physical component summary) ranges from 7.3 - 70.1; higher scores represent better functioning.
Time Frame: post-intervention survey
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Number analyzed (Participants) | 162 | 125 | 158 | 132
Score | 35.98 (10.05) | 38.01 (10.36) | 39.49 (11.70) | 36.18 (10.99)

8. Secondary Outcome: Hospitalization
Description: Hospitalization rates, measured as a total number of hospital admission for any reason per total patients year ("all-cause hospitalizations")
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: hospitalizations per patient year
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Number analyzed (Participants) | 377 | 342 | 401 | 286
hospitalizations per patient year | 1.55 [1.37 to 1.74] | 1.15 [0.098 to 1.32] | 1.37 [1.20 to 1.54] | 1.23 [1.04 to 1.42]

9. Primary Outcome: Dialysis Session Stability
Description: Systolic blood pressure (SBP) falling below 100 mmHg (using lowest SBP during session) if starting SBP ≥100.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: Proportion of sessions
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Number analyzed (Participants) | 377 | 342 | 401 | 286
Proportion of sessions | 0.202 (0.217) | 0.199 (0.204) | 0.172 (0.190) | 0.182 (0.205)

10. Secondary Outcome: Mortality
Description: Mortality rates, measured as a total number of deaths due to any cause per 100 patient years during the study period ("all-cause mortality").
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: Deaths per 100 patient years
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
Number analyzed (Participants) | 378 | 342 | 401 | 285
Deaths per 100 patient years | 16.99 [10.69 to 23.28] | 9.30 [4.43 to 14.17] | 14.85 [9.14 to 50.56] | 10.44 [4.76 to 16.11]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout all study periods: baseline (12 weeks), intervention (24 weeks), and follow up (12 weeks). Baseline monitoring was limited to counts of all-cause mortality because data for this time period were collected retrospectively.
Description: This was a pragmatic, low-risk trial with no changes to prescribed care. All-cause mortality was tracked. Adverse events relating to a breach in confidentiality were not observed. Other adverse events were not systematically tracked because the patient is very ill at baseline.
Arm/Group | No Intervention | Patient Activation | Provider Education | Patient and Provider
All-Cause Mortality (participants affected / at risk) | 45/382 | 30/346 | 35/410 | 27/293
Serious Adverse Events (participants affected / at risk) | 0/382 | 0/346 | 0/410 | 0/293
Other Adverse Events (participants affected / at risk) | 0/382 | 0/346 | 0/410 | 0/293

LIMITATIONS AND CAVEATS:
Results displayed for the primary and secondary outcomes are based on data from the 24-week intervention period, with the exception of quality of life measures based on the post-intervention quality of life survey conducted annually in each clinic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT03171545/Prot_SAP_000.pdf